CLINICAL TRIAL: NCT00138463
Title: Investigation of the Natural History of West Nile Virus Infection in Patients With Recently Acquired West Nile Fever or Neuroinvasive Disease
Brief Title: West Nile Virus Natural History
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Other Study IDs: 03-114; CASG 211; N01AI30025C; N01AI30025 (NIH)
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2010-02

CONDITIONS: West Nile Virus
Keywords: West Nile Virus, Neuroinvasive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, urine, serum.

GROUPS / COHORTS (2):
- West Nile Virus (WNV) Neuroinvasive Disease Cohort: Fever (temperature > 38 C) documented by a health care provider AND: at least one of the following, as documented by a health care provider and in the absence of a more likely clinical explanation: acutely altered mental status; other acute signs of central or peripheral neurologic dysfunction; or cerebrospinal fluid (CSF) pleocytosis associated with illness clinically compatible with meningitis.
- West Nile Virus Fever Cohort: Temperature > 38 C as documented by a health care provider.

SUMMARY:
West Nile Virus causes an infection that is spread to humans when bitten by certain types of mosquitoes. Mosquitoes become infected by biting infected birds. The purpose of this study is to find out more about West Nile Virus, which may assist in the design of better treatments. The study will be looking at the effects of the disease on individuals, specifically their nervous systems, and the outcomes of the disease. Study participants will include 120 adults ages 18 and older, who have either a fever and/or changes in their neurological (involving the brain and nervous system) status due to documented West Nile Virus infection. Study procedures will include physical examinations, blood tests, urine tests, cerebral spinal fluid (fluid in and around the brain and spinal cord) tests, and neurological (nervous system) testing. Study participants will be followed for 12 months.

DETAILED DESCRIPTION:
This is a multi-center, prospective, natural history study designed to characterize West Nile Virus (WNV) disease, including functional and neurologic outcomes, in study participants with laboratory documented WNV infection that have symptoms consistent with WNV neuroinvasive disease or WNV fever. The objectives of the study are to: identify and describe the mortality and morbidity, specifically neurologic and functional outcomes of patients with WNV; characterize the clinical course and diverse manifestations of WNV disease; and assess the kinetics of humoral immune responses to WNV infection, and to correlate these responses with clinical outcomes. The study will enroll a proposed sample size 120 study participants ages 18 and older. All study participants will undergo a series of laboratory, neurologic, and physical examinations and will be followed prospectively for one year to characterize the spectrum and sequelae of WNV disease. When patients meet inclusion criteria, informed consent will be obtained, and blood will be collected to perform polymerase chain reaction (PCR), immunoglobulin (Ig)M, and IgG testing for WNV infection. Urine PCR for WNV will also be obtained. Upon enrollment (Day 1), a medical and surgical history, review of systems, travel, vector and blood product history will be obtained, and the baseline neurologic and clinical status will be evaluated. A clinical assessment, including a physical examination, vital signs and laboratory assessment will be performed. Based on history a pre-illness neurologic functional score will be estimated, using the Barthel Index (BI) and the Modified Rankin Scale (MRS). Investigators will assess a Day 1 functional score, using the BI, the Modified Mini-Mental Status Examination (3MS), the Glasgow Outcome Score (GOS), and the Glasgow Coma Scale (GCS) if hospitalized and recorded answers to questions abstracted from the MRS on the day of entry into the study. At study visit Day 1 ± 3, cerebrospinal fluid (CSF) will be obtained and tested for cell count, differential, protein and glucose, IgM, IgG and PCR for WNV infection. If a study participant has a lumbar puncture conducted for standard of care at any time up to 72 hours prior and up to 72 hours after study enrollment, a repeat lumbar puncture will not be necessary if an adequate aliquot of CSF is available for shipment to the Collaborative Antiviral Study Group (CASG) Virology Laboratory and if the required cell count, differential, protein and glucose tests were performed. A brain Magnetic Resonance Imaging (MRI) scan will be done on study visit Day 1 ± 3. If the brain MRI scan on study visit Day 1 ± 3 suggests abnormalities, a repeat MRI scan will be conducted at study visit Day 30 ± 5. If changes (either improvement or worsening) in the WNV related lesions have occurred since the MRI conducted on study visit Day 1 ± 3, a third MRI will be conducted on study visit Day 90 ± 14. Subsequent MRIs will be conducted at study visits 180 ± 21 and 365 ± 30 only if the WNV related lesions continue to improve or worsen: any two MRIs where the WNV related lesions remain stable will obviate the need for further MRI scans. There will be study visits at Day 1, Day 14 ± 3, Day 30 ± 5, Day 90 ± 14, Day 180 ± 21, and Day 365 ± 30. At these visits a brief physical examination will be done, a functional score will be assigned, and blood will be obtained for serologic WNV studies. Neurological endpoints will include the GCS and 4 validated functional and cognitive scoring scales: The BI, MRS, GOS, and 3MS. MRI of spinal cord, electromyogram and nerve conduction studies will be included when available.

ELIGIBILITY:
Inclusion Criteria:

Patients, regardless of race or gender, who consent and meet entry criteria, will be enrolled.

* Greater than or equal to 18 years of age
* Documented West Nile Virus (WNV) infection (fever or neuroinvasive disease) that began within four months prior to study entry. Illness onset is defined as the first visit to a medical care provider where compatible symptoms (see cohort A and B below) are documented.
* Local laboratory documentation of WNV infection as defined by positive immunoglobulin (Ig) M and/or polymerase chain reaction (PCR) for WNV in serum or cerebrospinal fluid (CSF) concurrent with or following illness onset.
* Qualification for A or B Cohort.

Cohort A: Neuroinvasive Disease Cohort:

* Fever (temperature greater than 38 degrees Celsius) documented by a health care provider.
* AND: at least one of the following, as documented by a health care provider and in the absence of a more likely clinical explanation:

  1. Acutely altered mental status (e.g., disorientation, obtundation, stupor, or coma),
  2. Other acute signs of central or peripheral neurologic dysfunction (e.g., paresis or paralysis, nerve palsies, sensory deficits, abnormal reflexes, generalized convulsions, or abnormal movements), or
  3. CSF pleocytosis (white blood cell count greater than or equal to 4 per mm^3 corrected for red blood cell contamination in CSF) associated with illness clinically compatible with meningitis (e.g., headache or stiff neck).

     Cohort B: West Nile Virus Fever Cohort:
* Temperature greater than 38 degrees Celsius as documented by a health care provider.

Exclusion Criteria:

* Unable to obtain valid informed consent.
* Alternate explanation (as determined by the investigator) for clinical findings (such as structural brain lesion, cerebrovascular accident, or other infectious disease).
* Evidence of a microbial organism demonstrable on gram or fungal stain of cerebrospinal fluid (CSF) within four months prior to study entry.
* Investigator's opinion that patient would be unable to adhere to protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, 18 and older, all study participants must have been diagnosed with West Nile Virus (WNV) disease within the four months prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2003-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Identify and describe the mortality and morbidity, specifically neurologic and functional outcomes of patients with West Nile Virus disease. | Duration of Study.
Characterize the clinical course and diverse manifestations of West Nile Virus disease. | Duration of Study.
Assess the kinetics of humoral immune responses to West Nile Virus infection, and correlate these responses with clinical outcomes. | Analysis.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (27):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Kaiser Permanente South Bay Medical Center, Harbor City, California
  - University of Southern California, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Santa Rosa Kaiser Medical, Santa Rosa, California
  - Kaiser Permanente/Franklin Medical Center, Denver, Colorado
  - Idaho Falls Infectious Diseases, PLLC, Idaho Falls, Idaho
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health, Bethesda, Maryland
  - Saint Louis University, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Central Nebraska Medical Clinic, Broken Bow, Nebraska
  - VA Medical Center - Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. George University Clara Maas Medical Center, Belleville, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - University of Toledo, Toledo, Ohio
  - Memorial Hospital of RI, Pawtucket, Rhode Island
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas Health Science Center, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Hart J Jr, Tillman G, Kraut MA, Chiang HS, Strain JF, Li Y, Agrawal AG, Jester P, Gnann JW Jr, Whitley RJ; NIAID Collaborative Antiviral Study Group West Nile Virus 210 Protocol Team. West Nile virus neuroinvasive disease: neurological manifestations and prospective longitudinal outcomes. BMC Infect Dis. 2014 May 9;14:248. doi: 10.1186/1471-2334-14-248. PMID 24884681